CLINICAL TRIAL: NCT00551694
Title: A Second Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of a Single and a Repeat Oral Dose of GSK256073A in Healthy Adult Subjects
Brief Title: A Second Study to Determine the Effect of GSK256073A on HVTs
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HMA110541
Record Dates: First submitted 2007-10-29; First posted 2007-10-31 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2011-02

CONDITIONS: Healthy Subjects; Dyslipidaemias
Keywords: GSK256073A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GSK256073A tablets

SUMMARY:
The purpose of this study is to compare the effects of single and repeat doses of GSK256073 with placebo in HVT subjects that have been administrated GSK256073 in the HMA107787 study

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible physician, based on a medical evaluation including history, physical examination, laboratory tests, cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator considers that the finding will not introduce additional risk factors and will not interfere with the study procedures
* Healthy adult males or females between 18 and 55 years of age, inclusive.
* Female subjects must be of non-childbearing potential including pre-menopausal females with documented (medical report verification) hysterectomy or double oophorectomy or postmenopausal defined as 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy, or documented hysterectomy - tubal ligation is not sufficient
* Body weight > 50 kg (110 pounds) and body mass index (BMI) between 19 and 31 where:
* Subjects with QTc < 450 msec at screening (or QTc < 480 msec for subjects with Bundle Branch Block).
* A signed and dated written informed consent prior to admission to the study
* The subject is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions

Exclusion Criteria:

* Any clinically relevant abnormality identified on the screening medical assessment, laboratory examination or ECG
* Systolic blood pressure < 100 mmHg or ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg at the screening visit
* History of significant cardiac arrhythmias.
* Active peptic ulcer disease (PUD) and/or history of PUD
* Screening test positive for H. pylori at the screening visit
* History of gout and/or hyperuricemia
* A serum creatinine concentration above the reference range
* History of kidney stones
* PT and/or aPTT above the reference range
* History of recurrent indigestion, stomach upset or diarrhea
* Liver function tests (LFTs) or creatinine phosphokinase (CPK) above the normal reference range
* Positive HIV, Hepatitis B surface antigen or Hepatitis C antibody within 3 months of screening
* Positive urine drug and alcohol screen at screening or predose on Day 1 of each period
* History of alcohol consumption exceeding, on average, 7 drinks/week for women or 14 drinks/week for men (1 drink = 5 ounces of wine or 12 ounces of beer or 1.5 ounces of hard liquor) within 6 months of the first dose of study medication or a positive alcohol test at screening
* History of use of tobacco or nicotine containing products within 6 months of screening or a positive urine cotinine screen
* Use of antimicrobials, proton pump inhibitors and bismuth containing medications within 2 weeks prior to testing for H. pylori at Screening
* Use of prescription (including hormone replacement therapy) or non-prescription drugs and vitamins within 7 days or 5 half-lives (whichever is longer) prior to administration of study medication. Use of prescription antibiotics within 14 days prior to administration of study medication. An exception is acetaminophen which is allowed at doses of < 2g/day
* Use of dietary/herbal supplements including (but not limited to) St. John's wort, kava, ephedra (ma huang), gingko biloba, DHEA, yohimbe, saw palmetto, ginseng and red yeast rice within 14 days prior to treatment with study medication
* The subject has participated in a clinical trial and has received a drug or a new chemical entity within 30 days or 5 half-lives, or twice the duration of the biological effect of any drug(whichever is longer) prior to the first dose of current study medication
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation
* Consumption of grapefruit or grapefruit juice within 7 days prior to the first dose of study medication
* Donation of blood in excess of 500 mL within 56 days prior to dosing
* Unwillingness of male subjects to use a condom/spermicide, in addition to having their female partner use another form of contraception, such as an IUD, diaphragm with spermicide, oral contraceptives, injectable progesterone, subdermal implants or a tubal ligation, if engaging in sexual intercourse with a female partner who could become pregnant. This criterion must be followed from the time of the first dose of study medication until 84 days after the last dose of study medication
* Pregnant or nursing women
* History of other than rare (once yearly or less) flushing, particularly in perimenopausal women
* A hemoglobin A1c above the normal reference range and/or fasting blood glucose ≥100 mg/dL at the screening visit
* History of intra-ocular pathology, including but not limited to retinitis, uveitis, retinal detachment and macular edema

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2007-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
AEs, 12-Lead ECG, vital signs, nursing/physician observation, safety lab tests, flushing throughout the study. | throughout the study.
AUC and Cmax | throughout the study
Measures of accumulation ratios throughout the study (Ro, Rp, and Rs)[Period 2] | throughout the study

SECONDARY OUTCOMES:
Tmax, t½, Ae, and CLr , Cmax, ss, Ct, t½, Ae, CLr, and accumulation ratios throughout the study | throughout the study
PD response: NEFA and TG (6 and 24 hours post- dose), LDL, HDL, ApoA1, ApoA2, Apo B and Lp(a) on Days 1, 14, and 15. | Days 1, 14, and 15

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Minneapolis, Minnesota, United States